CLINICAL TRIAL: NCT06901999
Title: Efficacy and Safety of Methotrexate (MTX) or Thiotepa (for MTX-Intolerant Patients) Combined With R-CHOP and Orelabrutinib in the Treatment of Systemic DLBCL With Central Nervous System Involvement
Brief Title: Methotrexate or Thiotepa Combined With R-CHOP and Orelabrutinib in CNSL Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Prof, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNSL-WL-001
Record Dates: First submitted 2025-01-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: CNS Lymphoma
MeSH Terms: interventions — orelabrutinib; Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MTX or Thiotepa(for MTX-Intolerant Patients) Combined with R-CHOP and Orelabrutinib therapy group (Experimental): For DLBCL patients with central nervous system involvement, administer methotrexate (MTX) or thiotepa (for patients intolerant to MTX) combined with R-CHOP and orelabrutinib for six cycles, with each cycle lasting 21 days. Following the completion of induction therapy, proceed with consolidation therapy. If the patient undergoes autologous stem cell transplantation, maintain orelabrutinib for one year; if not, maintain orelabrutinib for two years unless disease progression or intolerable toxicity occurs.
  Interventions: Drug: Orelabrutinib; Drug: RCHOP+MTX or Thiotepa

INTERVENTIONS:
Drug: Orelabrutinib — 150 mg qd po. D1-21, 6 cycles, 21 days per cycle For patients continue transplant, maitaining for 1 year follow-up; otherwise maintaining during 2 years of follow-up，unless disease progression or intolerable toxicity occurs.
Drug: RCHOP+MTX or Thiotepa — rituximab: 375 mg/m2, D0; cyclophosphamide: 750 mg/m2, D1; doxorubicin: 50 mg/m2, D1; vincristine: 1.4 mg/m2, D1; prednisone: 100 mg, D1-5; MTX: 3.5 g/m2, D0; Thiotepa: 40 mg/m2, D3; Induction therapy, 6 cycles, 21 days a cycle

SUMMARY:
This study is designed as an open-label, prospective, single-arm, single-center trial aimed at evaluating the efficacy and safety of MTX or Thiotepa combined with Orelabrutinib and standard chemotherapy regimens in the treatment of DLBCL patients with central nervous system involvement.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the study and voluntarily sign the informed consent form.
* Age: 14-80 years.
* Expected survival of more than 3 months, as determined by the investigator.
* Pathologically or cytologically confirmed diffuse large B-cell lymphoma (DLBCL) of B-cell origin through pathology or flow cytometry.
* Central nervous system (CNS) involvement, confirmed by at least one of the following:

  1. Symptoms related to CNS involvement.
  2. Abnormal findings on imaging.
  3. Pathological evidence (positive cerebrospinal fluid cytology, positive brain lesion biopsy or positive cerebrospinal fluid ctDNA).
* Any non-hematologic toxicity related to prior treatments must have resolved to Grade 1 or normal levels (per NCI CTCAE Version 5.0), except for alopecia.
* Bone marrow and organ function must meet the following criteria (without blood transfusion, G-CSF administration, or pharmacological correction within 14 days prior to screening):

Bone marrow function:

1)Absolute neutrophil count (ANC) ≥ 1.0 × 10⁹/L. 2)Platelet count ≥ 50 × 10⁹/L. 3)Hemoglobin ≥ 60 g/L.

* Liver function:

  1. Total bilirubin ≤ 1.5 × ULN (≤ 3.0 × ULN if liver metastasis is present).
  2. AST and ALT ≤ 2.5 × ULN (≤ 5.0 × ULN if liver metastasis is present).
* Coagulation function:

International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN.

• Renal function: Serum creatinine ≤ 1.5 × ULN or estimated creatinine clearance rate ≥ 30 mL/min (calculated using the Cockcroft-Gault formula): Male: Cr (mL/min) = (140 - age) × weight (kg) / [72 × serum creatinine (mg/dL)]. Female: Cr (mL/min) = (140 - age) × weight (kg) / [85 × serum creatinine (mg/dL)].

* Women of childbearing potential (WOCBP) and men with reproductive potential must agree to use effective contraception during the study and for 3 months after discontinuing treatment.
* Good compliance, with willingness to adhere to visit schedules, dosing regimens, laboratory tests, and other study procedures.-

Exclusion Criteria:

* Contraindications to any of the drugs included in the treatment regimen.
* History of active liver disease, including viral or other hepatitis or liver cirrhosis (Hepatitis B is defined as HBV-DNA exceeding the upper limit of normal; active Hepatitis C is defined as seropositive for HCV antibodies, but patients with HCV-RNA negative results can be included).
* Human immunodeficiency virus (HIV) infection.
* Congestive heart failure classified as greater than NYHA Class II by the New York Heart Association; history of acute myocardial infarction, unstable angina, stroke, or transient ischemic attack within the past six months.
* Congenital long QT syndrome or QTc > 480 ms (Note: QTc must be calculated using Friederica's formula: QTcF = QT / (RR)^0.33).
* Pregnant or breastfeeding women, or those planning to become pregnant during the study.
* History of confirmed neurological or psychiatric disorders, or a history of substance abuse or drug addiction.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) | the end of Cycle 6 (up to approximately 24 weeks)
  The CR rate is defined as the percentage of participants with CR, on the basis of investigator assessments, according to 2014 Lugano criteria.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 2 years
  Progression-free survival was defined as the time from the date of first treatment until the date of the first documented day of disease progression or relapse, according to 2014 Lugano criteria, or death from any cause, whichever occurred first.
Overall Survival (OS) | up to approximately 4 years
  Overall survival is defined as the time from the date of first treatment to the date of death from any cause.
The Overall Response Rate (ORR) | the end of Cycle 6 (up to approximately 24 weeks)
  The ORR is defined as percentage of participants with overall response including complete response (CR) and partial response (PR), on the basis of investigator assessments, according to 2014 Lugano criteria.

IPD SHARING:
Plan to Share IPD: No